CLINICAL TRIAL: NCT01355640
Title: A Randomized Controlled Trial of Breast-feeding and/or Non-nutritive Sucking as Analgesia for Chinese Term Infants Receiving Heel Lance
Brief Title: Two Methods of Analgesia for Chinese Term Infants Receiving Heel Lance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Pingni, Lecturer, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S2006471
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Heel Pain Syndrome
Keywords: heel lance; pain; newborn
MeSH Terms: conditions — Pain | interventions — Lactation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- breast-feeding group (Experimental): Mothers console their babies by breast-feeding during heel lance.
  Interventions: Other: breast-feeding
- non-nutritive sucking (Experimental): Every mother was given a vacuum pacifier( the brand is "Goodbaby") to console her baby during heel lance.
  Interventions: Other: non-nutritive sucking
- control group (No Intervention): A research nurse also explained the study to the control group parents. Standard clinic procedure for infant injection was also implemented. Mothers in control group also lay on the side of the bed comfortably with their infants in their arms after the infants' soiled diapers were changed.

INTERVENTIONS:
Other: breast-feeding — Mothers lay on the side of the bed comfortably with their infants in their arms after the infants' soiled diapers were changed. Mothers breast-fed their babies. The study was initiated when the infants were observed to have a large amount of areola in their mouth, with flanged lips and active jaw movements. Then two minutes after the breast-feeding, an experienced technician began to do heel lance, heel lance was given by the same experienced technician.Mothers breast-fed their babies two minutes before, during and eight minutes after the heel lance. Throughout the whole procedure, mothers were encouraged to continue breast-feeding when the babies stopped sucking and/or began to cry.
  Other Names: non-pharmacological intervention
  Arms: breast-feeding group
Other: non-nutritive sucking — Mothers lay on the side of the bed comfortably with their infants in their arms after the infants' soiled diapers were changed. Each mother in this group was given a vacuum pacifier( the brand is "Goodbaby") to console her baby. Heel lance was given by the same experienced technician. The study was initiated when the infants can suck the pacifier and hold it by himself without others' help. This generally requires half or one minute. Then two minutes after non-nutritive sucking, an experienced technician began to do heel lance. Babies sucked the pacifier two minutes before, during and eight minutes after heel lance. Throughout the whole procedure, mothers were encouraged to continue non-nutritive sucking when the babies stopped sucking and/or began to cry.
  Other Names: non-pharmacological intervention
  Arms: non-nutritive sucking

SUMMARY:
1. The purpose of this study is to research and compare two sucking modes' effect(breast-feeding and non-nutritive sucking) and difference,hypothesis is that these two kinds of methods can decrease pain for Chinese term infants receiving heel stick.
2. A convenient sample of 90 neonates from a hospital in Beijing undergoing heel stick for Newborn Screening Program Blood Test were enrolled. They were randomized into three groups:

   * breast-feeding group
   * non-nutritive sucking group
   * control group
3. The results showed that:

   * Breast-feeding can reduce crying and grimace time, increase oxygen saturation.
   * Non-nutritive sucking can delay grimace's starting time, increase oxygen saturation.

DETAILED DESCRIPTION:
Untreated pain will also cause long term impact on newborns,Some scientists in foreign countries have done some research on rats, they found that if rats were exposed to pain for a long time, its nociception neural circuit's development will be harmed, and the pain threshold will be lowered. For newborns, untreated pain will cause hypalgesia when they are in puberty and hyperalgesia after adulthood. The experience of pain in infancy also affects the babies' later life after they grow up, it may cause emotional problems, minimal brain dysfunction, social intercourse defect and so on. So it is very important to find out useful interventions to decrease pain in newborns, considering the long term impact and side effect of medicine, it is seldom to use medical interventions to decrease pain. Non-pharmacological interventions become quite important. In foreign countries, there have been kinds of useful non-pharmacological interventions such as kangaroo care, breast-feeding, sucrose and non-nutritive sucking. While in China, there are massage, positioning, sucrose, music and kangaroo care that proved to be effective to decrease pain in newborns. The investigators find few reports about breastfeeding or non-nutritive sucking's effect of decreasing pain in term newborns. For breast-feeding, it includes the nursing mother who has consoling impact, hugging, attention transferring, taste, the breast milk contains tryptophane, which is the precursor of N-acetyl-5-O-T that can raise up the density of β-endorphin, β-endorphin has analgesic effect. For non-nutritive sucking, it also contains attention transferring. It is said that non-nutritive sucking can raise up the pain threshold through stimulating the oral tactile recipient, or promote the releasing of 5-HT that modulates pain. Non-nutritive sucking can also lower the sensitivity of peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

* Infants were considered to be eligible if they have been three days old who need to receive heel lance for blood sampling test for phenylketonuria (PKU), hyperbilirubinemia, thyroid hypofunction.
* Parents of infants who met the research criteria were invited to participate in the study.

Exclusion Criteria:

* Infants were excluded if they had a concurrent illness.
* Preterm babies, and babies who have received any operation after birth.
* Infant' mother who had a fever or some illness was excluded.
* Infants for whom an informed parental consent could not be obtained were also excluded.
* During the heel lance, the infants who need to receive two heel lances were also excluded.

Min Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
changes in heart rate value and oxygen saturation value,time length of grimacing and crying | 1 minute before heel lance and 8 minutes after heel lance, the duration of facial grimacing and crying, heart rate and oxygen saturation values at every 15 seconds.Time length of heart rate, oxygen saturation returned to baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Jingli Chen, Master, Study Director — Peking Union Medical College